CLINICAL TRIAL: NCT04124757
Title: The Impact of Deep Versus Standard Muscle Relaxation on Intra-operative Safety During Laparoscopic Surgery: a Multicenter Strategy Study
Brief Title: Impact of Deep Versus Standard Muscle Relaxation on Intra-operative Safety
Acronym: EURORELAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Martijn Boon, Prinicipal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P19.065
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Neuromuscular Blockade; Rocuronium; Anesthetics; Anesthesia Complication; Neuromuscular Blocking Agents; Surgery--Complications
Keywords: Laparoscopy
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard neuromuscular blockade (No Intervention): Subjects will receive regular rocuronium induction dose, followed by bolus foses of 10 mg in case of insufficient conditions
- Deep neuromuscular block (Experimental): Subjects will receive high dose rocuronium induction dose followed by continuous rocuronium administration, to achieve a depth of neuromuscular block of 1-2 twitches post tetanic count
  Interventions: Other: Deep neuromuscular block

INTERVENTIONS:
Other: Deep neuromuscular block — Deep neuromuscular block will be achieved with high dose rocuronium to achieve a depth of 1-2 twitches post tetanic count
  Other Names: High dose rocuronium
  Arms: Deep neuromuscular block

SUMMARY:
Muscle relaxants are routinely applied during anesthesia to facilitate endotracheal intubation and to improve surgical working conditions. Several investigations have shown that a deep neuromuscular block (NMB) improves the surgical working conditions over a moderate NMB and effectively precludes sudden deterioration of the surgical field. However, whether the improvement of surgical working conditions translates into less intra- and postoperative complications remains uncertain. Small prospective or retrospective studies shown an decrease of the incidence of intraoperative adverse events and postoperative complications after a deep NMB. There is a need to confirm these outcome data prospectively, in a large number of patients and clinics and during a variety of surgical procedures.

DETAILED DESCRIPTION:
Muscle relaxants are routinely applied during anesthesia to facilitate endotracheal intubation and to improve surgical working conditions. Several investigations have shown that a deep neuromuscular block (NMB) (post tetanic count (PTC) 1-2 twitches) improves the surgical working conditions over a moderate NMB (TOF count 1-3 twitches) and effectively precludes sudden deterioration of the surgical field. However, whether the improvement of surgical working conditions translates into less intra- and postoperative complications remains uncertain. A recent retrospective analysis of neuromuscular management during laparoscopic retroperitoneal surgery showed a reduced rate of unplanned 30 day readmissions when a deep NMB over a moderate NMB was applied (3.8% vs. 12.7%).In addition, a pooled analysis of 4 randomized controlled trials comparing different levels of intra-abdominal pressure and neuromuscular blockade during laparoscopic donor nephrectomy, showed a significant reduction in the incidence of intra-operative surgical complications from 12.6% with moderate NMB to 4.8% with deep NMB.

These previous observations were made in small prospective or retrospective studies. There is a need to confirm these outcome data prospectively, in a larger prospective trial for a variety of surgical procedures. We therefore propose a multi-center, randomized controlled trial, to study the effect of a deep NMB (PTC 1-2 twitches) versus standard NMB (single induction dose rocuronium) in a variety of laparoscopic surgical procedures on the incidence of intraoperative adverse events and postoperative outcome data.

In this study the effect of deep neuromuscular block compared to standard neuromuscular block on intra-operative adverse events during laparoscopic surgery using the CLASSIC score system is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic procedure with a complexity according to the BUPA classification for case complexity: 'MAJOR', 'MAJOR Plus or 'COMPLEX MAJOR'
* ASA (merican society of anesthesiologists) class I-III
* > 18 years of age
* Ability to give oral and written informed consent

Exclusion Criteria:

* Low or intermediate complexity laparoscopic procedures (BUPA 'SIMPLE' or 'INTER')
* Known or suspected neuromuscular disorders impairing neuromuscular function
* Allergies to muscle relaxants, anesthetics or narcotics mentioned in paragraph 5.2
* A (family) history of malignant hyperthermia
* Women who are or may be pregnant or are currently breast feeding
* Chronic use of any type of opioid or psychotropic drug
* Use of NSAID's shorter than 5 days before surgery
* Indication for rapid sequence induction
* Contra-indication for sugammadex use (e.g. known sugammadex allergy or Glomerular Filtration Rate <30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique van Velzen, PhD, Principal Investigator — LUMC
Locations (8):
- Université De Lorraine, Nancy, Meurthe-et-Moselle, France
- Istituto Nazionale Dei Tumori, Milan, Italy
- Netherlands (5):
  - RadboudUMC, Nijmegen, Gelderland
  - LUMC, Leiden, South Holland
  - Noordwest ziekenhuis groep, Alkmaar
  - Netherlands Cancer institute, Amsterdam
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
- Hospital Universitari I Politecnic La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Protocol and SAP will be published before start study. CSR will be reported after article publication in a peer reviewed journal.
Supporting Information: Study Protocol, SAP
Time Frame: Protocol and Statistical Analysis Plan will be published before start study. Clinical Study Report will be reported after article publication in a peer reviewed journal.
Access Criteria: To be declared

REFERENCES:
- [Background] Boon M, Martini C, Yang HK, Sen SS, Bevers R, Warle M, Aarts L, Niesters M, Dahan A. Impact of high- versus low-dose neuromuscular blocking agent administration on unplanned 30-day readmission rates in retroperitoneal laparoscopic surgery. PLoS One. 2018 May 23;13(5):e0197036. doi: 10.1371/journal.pone.0197036. eCollection 2018. PMID 29791482
- [Background] Torensma B, Martini CH, Boon M, Olofsen E, In 't Veld B, Liem RS, Knook MT, Swank DJ, Dahan A. Deep Neuromuscular Block Improves Surgical Conditions during Bariatric Surgery and Reduces Postoperative Pain: A Randomized Double Blind Controlled Trial. PLoS One. 2016 Dec 9;11(12):e0167907. doi: 10.1371/journal.pone.0167907. eCollection 2016. PMID 27936214
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Rosenthal R, Hoffmann H, Clavien PA, Bucher HC, Dell-Kuster S. Definition and Classification of Intraoperative Complications (CLASSIC): Delphi Study and Pilot Evaluation. World J Surg. 2015 Jul;39(7):1663-71. doi: 10.1007/s00268-015-3003-y. PMID 25665678
- [Background] Madsen MV, Scheppan S, Mork E, Kissmeyer P, Rosenberg J, Gatke MR. Influence of deep neuromuscular block on the surgeons assessment of surgical conditions during laparotomy: a randomized controlled double blinded trial with rocuronium and sugammadex. Br J Anaesth. 2017 Sep 1;119(3):435-442. doi: 10.1093/bja/aex241. PMID 28969327
- [Background] Ozdemir-van Brunschot DMD, Braat AE, van der Jagt MFP, Scheffer GJ, Martini CH, Langenhuijsen JF, Dam RE, Huurman VA, Lam D, d'Ancona FC, Dahan A, Warle MC. Deep neuromuscular blockade improves surgical conditions during low-pressure pneumoperitoneum laparoscopic donor nephrectomy. Surg Endosc. 2018 Jan;32(1):245-251. doi: 10.1007/s00464-017-5670-2. Epub 2017 Jun 22. PMID 28643056
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Derived] Honing M, Reijnders-Boerboom G, Dell-Kuster S, van Velzen M, Martini C, Valenza F, Proto P, Cambronero OD, Broens S, Panhuizen I, Roozekrans M, Fuchs-Buder T, Boon M, Dahan A, Warle M. The impact of deep versus standard neuromuscular block on intraoperative safety during laparoscopic surgery: an international multicenter randomized controlled double-blind strategy trial - EURO-RELAX TRIAL. Trials. 2021 Oct 26;22(1):744. doi: 10.1186/s13063-021-05638-2. PMID 34702332
- See also: Link to calculate comprehensive complication index — https://www.assessurgery.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Block
Started | 367 | 364
Completed | 365 | 363
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Block | Total
Number analyzed (Participants) | 362 | 361 | 723
Age, Continuous [Mean (Standard Deviation); unit: year] | 58.4 (13.7) | 58.0 (13.5) | 58.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 139 | 289
  Male | 212 | 222 | 434
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 362 | 361 | 723

OUTCOME MEASURES:

1. Primary Outcome: Classic Score>1
Description: The incidence of symptomatic intra-operative adverse events requiring intervention or treatment (ClassIntra®grade >1) during laparoscopic surgery in the standard of care versus the deep NMB group, as scored by the attending surgeon and anesthesiologist at the end of every procedure. A recent update of the ClassIntra®grade also involved intraoperative adverse events related to anesthesia [Gawria et al 2023]. This study will use both the original classic scoring, as well as an adapted version of the updated classic scoring system.
  The Classic score; classification of intraoperative complications, is a 6 point scale ranging from no complications (0) to fatal complications (5).
Time Frame: Day of surgery
Measure: Number; unit: participants
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Block
Number analyzed (Participants) | 361 | 362
participants | 66 | 54

2. Secondary Outcome: L-SRS (Leiden Surgical Rating Scale)
Description: To study the effect of deep neuromuscular block compared to standard neuromuscular block on peroperative surgical working conditions following the Leiden Surgical Rating scale (a 5 point scale, ranging from poor (1) to excellent (5) surgical conditions.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Block
Number analyzed (Participants) | 361 | 362
units on a scale | 4.6 (0.5) | 4.9 (0.3)

3. Secondary Outcome: 30 Day Post-operative Complications
Description: To study the effect of deep neuromuscular block compared to standard neuromuscular block on 30 day post-operative complications according the Clavien-Dindo score en Comprehensive Complication Index and unplanned readmissions
Time Frame: 30 postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Block
Number analyzed (Participants) | 361 | 362
Participants | 142 | 139

4. Secondary Outcome: Quality of Recovery (QoR)
Description: To study the effect of deep neuromuscular block compared to standard neuromuscular block on Quality of Recovery at post-operative day 1, 2 according to the Quality of Recovery-40
Time Frame: 2 postoperative days
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life (QoL)
Description: To study the effect of deep neuromuscular block compared to standard neuromuscular block on Quality of life at post-operative day 30 Short Form-36
Time Frame: 30 postoperative days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Block
All-Cause Mortality (participants affected / at risk) | 0/361 | 0/362
Serious Adverse Events (participants affected / at risk) | 24/361 | 23/362
Other Adverse Events (participants affected / at risk) | 65/361 | 51/362
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Neuromuscular Blockade (N=361) | Deep Neuromuscular Block (N=362)
Unplanned readmission (Surgical and medical procedures) | 24 | 23 — Unplanned readmission rate within 30days after surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Neuromuscular Blockade (N=361) | Deep Neuromuscular Block (N=362)
postoperative nausea vomiting (Gastrointestinal disorders) | 65 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT04124757/Prot_SAP_000.pdf